CLINICAL TRIAL: NCT01886911
Title: Neural Correlates of Video Game Based Training to Foster Mindfulness and Prosocial Skills in Adolescents
Brief Title: Games & Well-Being Study
Acronym: GWB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Davidson-GWB; Bill & Melinda Gates (Other Grant/Funding Number: Bill & Melinda Gates Foundation); Grant Number (Other Grant/Funding Number: opp1033728)
Record Dates: First submitted 2013-06-19; First posted 2013-06-26 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-06

CONDITIONS: Attentional Processing; Adolescent Behavior
Keywords: prosocial behavior; prosocial; attention training; attention; empathy; emotion recognition
MeSH Terms: conditions — Adolescent Behavior; Altruism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control for Attention Intervention (Active Comparator): Attentional Control Game is an active control group. We expect subjects in this group to play a control game for 2 weeks (plus or minus 7 days).
  Interventions: Other: Control for Attention Intervention
- Prosocial Training Intervention Game (Experimental): The prosocial intervention group, which we expect will be play the experimental prosocial training game for 2 weeks (plus or minus 7 days).
  Interventions: Other: Prosocial Training Intervention Game
- Attention Training Intervention Game (Experimental): The attention intervention group, which we expect will be play the experimental attention training game for 2 weeks (plus or minus 7 days).
  Interventions: Other: Attention Training Intervention Game
- Control for Prosocial Intervention (Active Comparator): This is an active control group. We expect subjects in this group to play a control game for 2 weeks (plus or minus 7 days).
  Interventions: Other: Control for Prosocial Intervention

INTERVENTIONS:
Other: Attention Training Intervention Game
  Other Names: Tenacity
  Arms: Attention Training Intervention Game
Other: Prosocial Training Intervention Game
  Other Names: Crystals of Kaydor
  Arms: Prosocial Training Intervention Game
Other: Control for Attention Intervention
  Arms: Control for Attention Intervention
Other: Control for Prosocial Intervention
  Arms: Control for Prosocial Intervention

SUMMARY:
This project is focused on the neural and behavioral correlates of two different videos games that will be used as training tools. The two video games, developed by the Games Learning Society research group at the University of Wisconsin-Madison (UW) and the Wisconsin Institute for Discovery, are tailored to train mindfulness, particularly the regulation of attention; and prosocial behavior, especially sensitivity to others, in adolescents. This study will evaluate the hypothesis that systematic playing of mindfulness and prosocial games will change brain function in specific attentional, social and emotional circuits in potentially beneficial ways, and will impact performance on cognitive tasks of attention, and on measures of social cue perception and the propensity to share and behave altruistically. The investigators will employ behavioral and functional MRI-based neuroimaging measures to evaluate the investigators hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speaker
* Enrolled in 7th or 8th grade

Exclusion Criteria:

* Currently on psychotropic medications

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in behavioral measures | baseline and up to 3 weeks
  Change in behavioral measures before and after attentional video game training. Timeframe is up to 7 days following the end of the 2 week game playing period.
Change from baseline in fMRI | baseline and up to 3 weeks
  Change in fMRI neural markers of empathic accuracy before and after attentional video game training. Timeframe is up to 7 days following the 2 week game playing period.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Davidson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Patsenko EG, Adluru N, Birn RM, Stodola DE, Kral TRA, Farajian R, Flook L, Burghy CA, Steinkuehler C, Davidson RJ. Mindfulness video game improves connectivity of the fronto-parietal attentional network in adolescents: A multi-modal imaging study. Sci Rep. 2019 Dec 10;9(1):18667. doi: 10.1038/s41598-019-53393-x. PMID 31822684